CLINICAL TRIAL: NCT01016665
Title: Anastrozole Reduced Proliferation and Progesterone Receptor Indexes in Short Term Hormone Therapy. A Prospective Placebo Double Blind Study
Brief Title: Anastrozole Reduced Proliferation and Progesterone Receptor Indexes in Short Term Hormone Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Andre Mattar MD, Federal University of Sao Paulo
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: 0904/04
Record Dates: First submitted 2009-11-17; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Short Term; Homontherapy; aromatase inhibitor; Short term hormonetherapy in breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Anastrozole
- Tamoxifen (Other): Tamoxifen 20 mg day 26 days
  Interventions: Drug: Anastrozole
- Anastrozole (Other): Anastrozole 1mg 26 days
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — Tamoxifen 20mg and anastrozole 1 mg

SUMMARY:
Background: Identification of new biomarkers with potential predictive and prognostic role has contributed unequivocally to breast cancer treatment.

Although traditionally endocrine therapy is based on hormonal receptors status (estrogen - ER and progesterone- PR), some patients become hormone resistant. In order to identify a possible profile associated to hormonal resistance, some biomarkers have been assessed after short period primary hormone therapy (HT).

Objectives: To compare the expression of Ki-67, Bcl2, Bax, Bak, ER and e PR in postmenopausal women with ER positive invasive ductal carcinomas (IDC), prior and after tamoxifen and anastrozole in short term hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer post-menopausal women
* Estrogen and/or progesterone receptor positive

Exclusion Criteria:

* Patients with endocrine disease
* Hormone therapy users or those who had been pregnant in the last 12 months before the diagnosis
* Patients with a negative expression for estrogen and/or progesterone receptors
* Women with a history of thromboembolism
* Patients who had previously undergone any treatment for breast cancer

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Expression of progesterone | end of the study (june 2008)

SECONDARY OUTCOMES:
Expression of Ki-67 | end of the study (june 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Mattar, MD, Principal Investigator
Locations (1):
- Sao Paulo Federal University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Cuzick J, Powles T, Veronesi U, Forbes J, Edwards R, Ashley S, Boyle P. Overview of the main outcomes in breast-cancer prevention trials. Lancet. 2003 Jan 25;361(9354):296-300. doi: 10.1016/S0140-6736(03)12342-2. PMID 12559863
- [Result] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Result] Macaskill EJ, Renshaw L, Dixon JM. Neoadjuvant use of hormonal therapy in elderly patients with early or locally advanced hormone receptor-positive breast cancer. Oncologist. 2006 Nov-Dec;11(10):1081-8. doi: 10.1634/theoncologist.11-10-1081. PMID 17110627
- [Result] Dowsett M. Preoperative models to evaluate endocrine strategies for breast cancer. Clin Cancer Res. 2003 Jan;9(1 Pt 2):502S-10S. PMID 12538507
- [Result] Dixon JM, Renshaw L, Bellamy C, Stuart M, Hoctin-Boes G, Miller WR. The effects of neoadjuvant anastrozole (Arimidex) on tumor volume in postmenopausal women with breast cancer: a randomized, double-blind, single-center study. Clin Cancer Res. 2000 Jun;6(6):2229-35. PMID 10873072
- [Result] Harvey JM, Clark GM, Osborne CK, Allred DC. Estrogen receptor status by immunohistochemistry is superior to the ligand-binding assay for predicting response to adjuvant endocrine therapy in breast cancer. J Clin Oncol. 1999 May;17(5):1474-81. doi: 10.1200/JCO.1999.17.5.1474. PMID 10334533
- [Result] Musgrove EA, Sutherland RL. Biological determinants of endocrine resistance in breast cancer. Nat Rev Cancer. 2009 Sep;9(9):631-43. doi: 10.1038/nrc2713. PMID 19701242
- [Result] Miller WR, Dixon JM, Cameron DA, Anderson TJ. Biological and clinical effects of aromatase inhibitors in neoadjuvant therapy. J Steroid Biochem Mol Biol. 2001 Dec;79(1-5):103-7. doi: 10.1016/s0960-0760(01)00149-2. PMID 11850213
- [Result] Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, Griffith C, Boeddinghaus I, Salter J, Detre S, Hills M, Ashley S, Francis S, Walsh G, A'Hern R. Proliferation and apoptosis as markers of benefit in neoadjuvant endocrine therapy of breast cancer. Clin Cancer Res. 2006 Feb 1;12(3 Pt 2):1024s-1030s. doi: 10.1158/1078-0432.CCR-05-2127. PMID 16467120
- [Result] Konstantinidou AE, Korkolopoulou P, Patsouris E. Apoptotic markers for tumor recurrence: a minireview. Apoptosis. 2002 Oct;7(5):461-70. doi: 10.1023/a:1020091226673. PMID 12207179
- [Result] Ellis MJ, Tao Y, Luo J, A'Hern R, Evans DB, Bhatnagar AS, Chaudri Ross HA, von Kameke A, Miller WR, Smith I, Eiermann W, Dowsett M. Outcome prediction for estrogen receptor-positive breast cancer based on postneoadjuvant endocrine therapy tumor characteristics. J Natl Cancer Inst. 2008 Oct 1;100(19):1380-8. doi: 10.1093/jnci/djn309. Epub 2008 Sep 23. PMID 18812550
- [Result] Colozza M, Azambuja E, Cardoso F, Sotiriou C, Larsimont D, Piccart MJ. Proliferative markers as prognostic and predictive tools in early breast cancer: where are we now? Ann Oncol. 2005 Nov;16(11):1723-39. doi: 10.1093/annonc/mdi352. Epub 2005 Jun 24. PMID 15980158
- [Result] Dowsett M. Biomarker investigations from the ATAC trial: the role of TA01. Breast Cancer Res Treat. 2004;87 Suppl 1:S11-8. doi: 10.1007/s10549-004-1578-3. PMID 15597216
- [Result] Dowsett M, Ebbs SR, Dixon JM, Skene A, Griffith C, Boeddinghaus I, Salter J, Detre S, Hills M, Ashley S, Francis S, Walsh G, Smith IE. Biomarker changes during neoadjuvant anastrozole, tamoxifen, or the combination: influence of hormonal status and HER-2 in breast cancer--a study from the IMPACT trialists. J Clin Oncol. 2005 Apr 10;23(11):2477-92. doi: 10.1200/JCO.2005.07.559. Epub 2005 Mar 14. PMID 15767642
- [Result] Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, Griffith C, Boeddinghaus I, Salter J, Detre S, Hills M, Ashley S, Francis S, Walsh G; IMPACT Trialists. Short-term changes in Ki-67 during neoadjuvant treatment of primary breast cancer with anastrozole or tamoxifen alone or combined correlate with recurrence-free survival. Clin Cancer Res. 2005 Jan 15;11(2 Pt 2):951s-8s. PMID 15701892
- [Result] Ellis MJ, Ma C. Letrozole in the neoadjuvant setting: the P024 trial. Breast Cancer Res Treat. 2007;105 Suppl 1(Suppl 1):33-43. doi: 10.1007/s10549-007-9701-x. Epub 2007 Oct 3. PMID 17912634